CLINICAL TRIAL: NCT05474352
Title: Use of Water Warming/Cooling Garment to Maintain a Constant Intraoperative Core Target Temperature in Patients Undergoing Cytoreductive Surgery With Hyperthermic Intraperitoneal Chemotherapy (HIPEC): A Proof-of-Concept Study
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: 0 participants enrolled
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-0159; NCI-2022-05348 (Other: NCI CTRP-Clinical Trials Reporting Registry)
Record Dates: First submitted 2022-06-20; First posted 2022-07-26 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Hyperthermic Intraperitoneal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- ALLON System (Experimental): The ALLON system water garment, is like a large apron that covers your body. There are tubes that run throughout the water garment, which allow warm liquid to flow so that the garment keeps the participant warm. The ALLON system water garment will be filled with warm water.
  Interventions: Device: Allon System

INTERVENTIONS:
Device: Allon System — Water garments (Allon system) already pre-filled with warm water will be set up before induction of anesthesia. After the induction of general anesthesia, the water garment will cover the lower and upper extremities, the lateral portion of the chest, and the entire back of the patient, which accounts for 70% of the body surface. The water garment will be opened temporarily on the upper extremities for intravenous access and arterial line placement and will be continued intraoperatively until the patient is transferred from the OR table to the stretcher

SUMMARY:
To look at the feasibility of using a water warming/cooling garment (called the ALLON system) to maintain a target body temperature during surgery and chemotherapy perfusion (a method of pouring chemotherapy throughout your abdominal cavity) without overheating or overcooling your body.

DETAILED DESCRIPTION:
Objectives:

Primary Objectives:

To evaluate the feasibility of using a water warming/cooling garment (Allon system) to achieve and maintain a bladder temperature of ≥38°C for at least 30 minutes or longer during cytoreductive surgery with hyperthermic intraperitoneal chemotherapy while avoiding core (esophageal) hyperthermia (≥39.5°C).

Secondary Objective:

To evaluate the safety for all study participants when using of the Allon system strategy in achieving and maintaining a bladder temperature of ≥38°C for at least 30 minutes or longer during cytoreductive surgery with hyperthermic intraperitoneal chemotherapy while avoiding core hyperthermia (≥39°C)

ELIGIBILITY:
Inclusion Criteria:

* Adults patients (>18 years old)
* Cytoreductive surgery with hyperthermic intraperitoneal chemotherapy with an expected duration of perfusion longer than 60 minutes
* Signed informed consent

Exclusion criteria:

* America Society of Anesthesiology (ASA)physical status >4
* Patient undergoing cytoreductive surgery with hyperthermic intraperitoneal chemotherapy for recurrent disease.
* Patients with open wounds
* Patients with a history of thermoregulatory diseases such as spinal cord injury, thyroid disease, and malignant hyperthermia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
Number of Patients to achieve and maintain a bladder temperature of ≥38°C for at least 30 minutes or longer. | through HIPEC surgery (up to 4 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Maria F Ramirez, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org